CLINICAL TRIAL: NCT03478618
Title: Comparison of Two Different Protocols of Fluid Therapy in Severe Preeclamptic Patients Under Spinal Anesthesia : Hemodynamic and Kidney Function Outcome
Brief Title: Comparison of Different Protocols of Fluid Therapy in Severe Preeclamptic Patients Under Spinal Anesthesia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Bola Fawzi Mekhail Sedrak, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: haemodynamics in preeclampsia
Record Dates: First submitted 2018-03-21; First posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Hypotension Drug-Induced
MeSH Terms: conditions — Hypotension | interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group R (Active Comparator): 30 patients will receive 15ml/kg/h lactated Ringer (LR) intraoperative.
  Interventions: Drug: Lactated Ringer
- Group L (Active Comparator): 30 patients will receive 30ml/kg/h lactated Ringer (LR) intraoperative.
  Interventions: Drug: Lactated Ringer

INTERVENTIONS:
Drug: Lactated Ringer — Patients will be divided into 2 groups according to the amount of fluids received during caesarian section under spinal anesthesia.
  Group (R) 30 patients will receive 15ml/kg/h lactated Ringer (LR) intraoperative. Group (L) 30 patients will receive 30ml/kg/h lactated Ringer (LR) intraoperative. blood loss will be replaced if more than 500 ml in ratio 3 ml crystalloid : 1ml blood in both groups

SUMMARY:
To compare the effect of two different protocol of fluid therapy in sever preeclamptic patients under spinal anesthesia : Hemodynamic and kidney function .

ELIGIBILITY:
Inclusion Criteria:

* more than 36 weeks gestation
* singleton pregnant women planned for elective caesarian section

Exclusion Criteria:

* patient refusal.
* psychiatric disorders.
* parturient <36 weeks gestation, twins, abnormal cardiotocography (CTG) tracing.
* absolute contraindications for spinal anesthesia (patients refusal, raised intracranial pressure, hypovolemic states, abnormal coagulopathy).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
incidence of hypotension | 1 hour
  decrease in systolic blood pressure more than 20% of base line

REFERENCES:
- [Background] Ansari MR, Laghari MS, Solangi KB. Acute renal failure in pregnancy: one year observational study at Liaquat University Hospital, Hyderabad. J Pak Med Assoc. 2008 Feb;58(2):61-4. PMID 18333521
- [Background] Ganesan C, Maynard SE. Acute kidney injury in pregnancy: the thrombotic microangiopathies. J Nephrol. 2011 Sep-Oct;24(5):554-63. doi: 10.5301/JN.2011.6250. PMID 21240869